CLINICAL TRIAL: NCT03378739
Title: Implementation of a Cardiogenic Shock Team and Clinical Outcomes (INOVA-SHOCK Registry)
Brief Title: Inova Cardiogenic Shock Registry (INOVA SHOCK)
Acronym: INOVASHOCK
Status: Recruiting | Type: Observational
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Other Study IDs: 172870
Record Dates: First submitted 2017-12-12; First posted 2017-12-20 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cardiogenic Shock
Keywords: cardiogenic; shock
MeSH Terms: conditions — Shock, Cardiogenic; Shock

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiogenic Shock team activation — Any patient with cardiogenic shock, whether inpatient or transferred from another facility, treated at the Inova Heart and Vascular Institute by the designated Cardiogenic Shock Team.

SUMMARY:
To collect retrospective clinical outcomes related to acute decompensated heart failure cardiogenic shock, acute myocardial infarction cardiogenic shock and compare current versus historical survival rates.

To collect Inova Heart and Vascular Institute (IHVI) site specific outcomes before and after initiation of the Cardiogenic Shock team on January 1, 2017.

To collect outcomes related to implementation of mechanical circulatory support versus no circulatory intervention and type of intervention (extracorporeal membrane oxygenation (ECMO) versus intracorporeal axial-flow (Impella).

• Assess survival at three time points.

DETAILED DESCRIPTION:
Any patient with cardiogenic shock, whether inpatient or transferred from another facility, treated at the Inova Heart and Vascular Institute shall be included in this registry. This includes adults with and without decision making capacity over the age of 18 years old.

The primary investigator (PI) will designate the data points to be included in the database in order to assess the efficiency of procedures and protocols in the treatment of cardiogenic shock at the IHVI as administered by the Shock team, to identify relationships between treatment and negative morbidity and mortality outcomes, and to monitor and improve quality of care delivered.

ELIGIBILITY:
Inclusion Criteria:

-Patients at the IHVI with documented Cardiogenic Shock team intervention for acute decompensated heart failure cardiogenic shock, or acute myocardial infarction cardiogenic shock.

Exclusion Criteria:

-Patients under the age of 18 will be excluded.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients at the IHVI with documented Cardiogenic Shock team intervention for acute decompensated heart failure cardiogenic shock, or acute myocardial infarction cardiogenic shock
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective review of Cardiogenic shock patients outcomes | 1 Year
  To create an archive of retrospective clinical outcomes (acute decompensated heart failure cardiogenic shock, or acute myocardial infarction cardiogenic shock) and compare current versus historical survival rates.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Truesdell, MD, Principal Investigator — Inova Health Care Services; Behnam Tehrani, MD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
To facilitate both national and international research efforts in cardiogenic shock patient's collaborative studies may occur with other institutions outside of Inova.
Supporting Information: CSR

REFERENCES:
- [Derived] Sinha SS, Rosner CM, Tehrani BN, Maini A, Truesdell AG, Lee SB, Bagchi P, Cameron J, Damluji AA, Desai M, Desai SS, Epps KC, deFilippi C, Flanagan MC, Genovese L, Moukhachen H, Park JJ, Psotka MA, Raja A, Shah P, Sherwood MW, Singh R, Tang D, Young KD, Welch T, O'Connor CM, Batchelor WB. Cardiogenic Shock From Heart Failure Versus Acute Myocardial Infarction: Clinical Characteristics, Hospital Course, and 1-Year Outcomes. Circ Heart Fail. 2022 Jun;15(6):e009279. doi: 10.1161/CIRCHEARTFAILURE.121.009279. Epub 2022 May 5. PMID 35510546
- [Derived] Tehrani B, Truesdell A, Singh R, Murphy C, Saulino P. Implementation of a Cardiogenic Shock Team and Clinical Outcomes (INOVA-SHOCK Registry): Observational and Retrospective Study. JMIR Res Protoc. 2018 Jun 28;7(6):e160. doi: 10.2196/resprot.9761. PMID 29954728